CLINICAL TRIAL: NCT05451394
Title: Prevention of Fall Injury in Military Settings Through the Use of Body Awareness.
Brief Title: Prevention of Injury in Military Settings Through the Use of Body Awareness.
Acronym: POSITION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2020PBMD04
Record Dates: First submitted 2021-10-14; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Traumatic Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The preventive program will be deployed in the first unit selection camp, then in the second the "active control program" will be deployed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROAF Arm (Experimental): 6 one-hour workshops working on enhancing postural awareness through the use of ROAF
  Interventions: Other: ROAF
- Active control (Active Comparator): 6 one-hour workshops on higher cognitive processes (memory, attention...)
  Interventions: Other: Active Comparator

INTERVENTIONS:
Other: ROAF — Use of the method "Ressource Optimisation of Armed Forces (ROAF). 6 one-hour workshops
  Arms: ROAF Arm
Other: Active Comparator — 6 one-hour workshops on cognitive process
  Arms: Active control

SUMMARY:
The POSITION project aims to investigate the cognitive mechanism of postural body awareness as a risk factor for injury and as a target for a primary prevention strategy based on the Resource Optimization of Armed Forces (ROAF) method.

DETAILED DESCRIPTION:
Physical activity and sport play an important role in the military environment to develop and optimize the operational capability of warfighters. Nevertheless, the prevalence of injuries is high and the identification of risk factors accessible to primary prevention measures is a major challenge for the protection of warfighter health. Military epidemiologic data show that the majority of injuries are acute fall-type injuries following a loss of balance. These data suggest that the quality of postural balance may influence the occurrence of injuries encountered during military physical activities. The high level of stress to which individuals are exposed during military physical activities could contribute to the degradation of postural balance quality. The POSITION project aims to study the cognitive mechanism of postural body awareness as a risk factor for injury and as a target for a primary prevention strategy based on the Resource Optimization of Armed Forces (ROAF) method. ROAF could improve postural control and decrease the intensity of the psychobiological stress response, and thus reduce the incidence rate of fall injuries occurring during military physical activities.

ELIGIBILITY:
Inclusion Criteria:

* Signing an informed consent to participate in the study
* enrolled in the selection camp
* Be affiliated to a Social Security system

Exclusion Criteria:

* advanced ROAF formation (over 10 hours)
* Refusal to participate
* Person covered by articles L1121-5 to L1121-8 of the public health code, namely

  * Pregnant women, women in labour or nursing mothers,
  * person deprived of liberty by judicial or administrative decision,
  * persons subject to psychiatric monitoring under Articles L3112-1 and L3113-1 who are not covered by the provisions of Article L1121-8,
  * adult persons who are subject to a legal protection measure or who are unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-10-17 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of imbalance injuries in each of the two groups (ROAF vs active control). | 3 weeks
  The primary endpoint will be the incidence rate of imbalance injuries in each of the two groups (ROAF vs active control).

SECONDARY OUTCOMES:
Evolution of postural awareness measured by the postural awareness scale. | 3 weeks
  Evolution of the self-questionnaire measuring postural awareness completed at inclusion, at the final visit and at the beginning of each workshop; 8 times in total.
Evolution of postural balance | 3 weeks
  Difference between postural balance assessed during the inclusion visit and the final visit, using a posturography tool.
Evolution of the stress level measured by the perceived stress scale | 3 weeks
  Evolution of the self-questionnaire measuring perceived stress completed at inclusion, at the final visit, and at the beginning of each workshop; 8 times in total.
Evolution of the hormonal stress level. | 3 weeks
  Difference of levels of hormonal stress in a saliva sample (at the inclusion and final visit).

CONTACTS AND LOCATIONS:
Locations (1):
- French Army, Paris, France

REFERENCES:
- [Derived] Obligi L, Bertrand M, Boivent M, Corcostegui SP, Coz PE, Derkenne C, Des Robert V, Hurpin V, Hus J, L'Hermitte B, Lely L, Patey E, Romary E, Saint-Jean L, Trente A, Turpin M, Vertu N, Verdonk C, Duffaud AM. Position: A study protocol for the prevention of fall injuries in french special forces selection courses using a body-centered intervention. PLoS One. 2023 Oct 4;18(10):e0290241. doi: 10.1371/journal.pone.0290241. eCollection 2023. PMID 37792797